CLINICAL TRIAL: NCT02962921
Title: Acute Insulin Effects on Cardiac Function in Patients With Diabetes Mellitus
Brief Title: Insulin Effects on Cardiac Function in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1558-RMB-CTIL
Record Dates: First submitted 2016-09-10; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus; Ventricular Dysfunction
MeSH Terms: conditions — Diabetes Mellitus; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetic patients (Experimental): Diabetic patients were treated with insulin loads, left ventricle functional parameters were compared to those of healthy persons.
  Metabolic indices of insulin effect: blood insulin levels, glucose disposal rates under insulin infusion, were compared to respective group of healthy persons, studied earlier at our institution Insulin LISPRO intravenous loading
  Interventions: Drug: Insulin LISPRO intravenous loading

INTERVENTIONS:
Drug: Insulin LISPRO intravenous loading — intravenous infusion of insulin Lispro.
  Other Names: Humalog Insulin

SUMMARY:
Our investigation studies the role of acute insulin administration on the diabetic heart, its corresponding effective blood-insulin level and the time-course applicability of insulin in a routine clinical setting.

A case series of six male (48.1 ± 4.9 y/o) patients with controlled diabetes (HbA1c of 6.6 ± 0.3%, disease duration of 14.4 ± 6.7 yr). Each subject was evaluated for glucose homeostatic, hemodynamic and echocardiographic systolic and diastolic parameters at baseline and following two successive insulin-load steps of a euglycemic hyperinsulinemic clamp study, each 2 h in duration. Results are presented as a mean ± SEM and analysed using the student's t-test.

DETAILED DESCRIPTION:
Patients:

Six male diabetic (five type 2 and one type 1) patients, 30-65 year old, with an established diagnosis of diabetes mellitus for ≥2 years, who were free of significant valvular heart disease, atrial arrhythmia or cardiac pacing comprised the study population. Patients' characteristics are summarized in table 1.

Each patient served as his or her own control. The study protocol was approved by the ethics committee at Rambam Medical Center, Haifa, Israel. Prior to the study, patients gave written informed consent after receiving a detailed explanation as to the purpose of the study, the technique, its side effects and the study protocol.

Patients were studied within a clinical research facility at the Rambam Medical Center, Haifa, Israel. Baseline evaluation was conducted at 8:00 am after 12 h of fasting, followed by two hyperinsulinemic euglycemic clamp (EHC) steps (2 h each step); The following vital signs were monitored during the study protocol: manual heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP) and baseline 12-lead electrocardiogram (ECG) recording. Glucose consumption rates against changing insulin levels were measured by the EHC technique. Cardiac function parameters were measured in the last 10 min of each step by tissue Doppler echocardiography. Results are presented as a mean ± SEM.

Clamp technique:

Each patient underwent an EHC study according to the protocol described previously, and implemented in our institute. Baseline measurements of blood insulin and glucose levels were collected. Thereafter, two insulin loads were initiated. The blood glucose level was kept near euglycemia (90 ± 5 mg/dl) throughout 2 h period of each insulin load step. Intravenous (iv) insulin loads were administered by 1- and 10-mU/kg·min at steps 1 and 2 of insulin loading (Lispro Insulin, Eli Lilly, France), respectively. Dexstrose in water 50% (DW50) was infused at variable infusion rates, titrated to maintain euglycemia. Concomitant saline 0.45% was used to dilute the DW50 in order to prevent hypertonicity-induced irritation of the cannuled vein. During the baseline period, saline 0.45% infusion rates were 0.75 ml/min to keep the iv cannule open. Every patient was given a chance to urinate before step 2.

Glucose and insulin homeostatic parameters of the study group were compared to those of healthy controls we studied earlier.

Cardiac function assessment:

Transthoracic echocardiography was performed by a qualified echocardiographer using a General Electric Vivid 3 machine (Tirat HaCarmel, Israel). Parameters were assessed as the mean of three consecutive heart beats.

Systolic echocardiographic parameters:

LV fractional shortening (LVFS) derived from end diastolic and end systolic LV dimensions; LV ejection fraction (LVEF) derived from end diastolic and end systolic LV volumes.

Diastolic echocardiographic parameters:

1. Mitral valve diastolic flow parameters by pulse wave Doppler: E wave, represents early diastolic filling; A wave, represents late diastolic filling concomitant with the atrial kick, E/A ratio and E wave deceleration time (DT).
2. Tissue Doppler-derived velocities of the mitral annulus: E' represents early diastolic velocity synchronous to the mitral inflow E wave, measured close to the interventricular septum (E' medial) and lateral wall (E' lateral); E' mean, derived from E' lateral and E' medial. A' represents late diastolic velocity to the synchronous mitral inflow A wave, measured close to the septum (A' medial) and lateral wall (A' lateral). A' mean is derived from A' lat. and A' med. A' reflects mitral annulus movement during atrial contraction. The E to E' ratio represents diastolic LV compliance.

Results are presented as mean ± SEM and analyzed using the student's t-test. Statistical significance considered when p value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus duration of 2 years and over.

Exclusion Criteria:

* Previous cardiac disease: valvular, Pacing, Arrhythmias, Primary Cardiomyopathy.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-02; Primary Completion 2003-05 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Left ventricle ejection fraction (%) | 1 year

SECONDARY OUTCOMES:
Time needed to exert insulin effect on myocardial function (hour) | 1 year
  Describe the shortest time required for insulin to change myocardial function.

OTHER OUTCOMES:
Blood insulin levels (μU/ml: micro international unit per milliliter) | 1 year
Left ventricle fractioning shortening (%) | 1 year
E wave (centimeter per second) | 1 year
A wave (centimeter per second) | 1 year
E deceleration time (seconds) | 1 year
E' (centimeters) | 1 year
A' (centimeters) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Karnieli, MD, Study Chair — Professor emeritus, Faculty of medicine, Technion. Haifa, Israel; Ronen Bar Yoseph, MD, Principal Investigator — Pediatric Pulmonary Institute; Sergey Yalonetsky, MD, Principal Investigator — Cardiology Division
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
First we need to learn how to share data

REFERENCES:
- [Result] Adeghate E. Molecular and cellular basis of the aetiology and management of diabetic cardiomyopathy: a short review. Mol Cell Biochem. 2004 Jun;261(1-2):187-91. doi: 10.1023/b:mcbi.0000028755.86521.11. PMID 15362503
- [Result] Francis GS. Diabetic cardiomyopathy: fact or fiction? Heart. 2001 Mar;85(3):247-8. doi: 10.1136/heart.85.3.247. No abstract available. PMID 11179253
- [Result] Kitzman DW, Gardin JM, Gottdiener JS, Arnold A, Boineau R, Aurigemma G, Marino EK, Lyles M, Cushman M, Enright PL; Cardiovascular Health Study Research Group. Importance of heart failure with preserved systolic function in patients > or = 65 years of age. CHS Research Group. Cardiovascular Health Study. Am J Cardiol. 2001 Feb 15;87(4):413-9. doi: 10.1016/s0002-9149(00)01393-x. PMID 11179524
- [Result] Gutierrez C, Blanchard DG. Diastolic heart failure: challenges of diagnosis and treatment. Am Fam Physician. 2004 Jun 1;69(11):2609-16. PMID 15202695
- [Result] McMurray JJ, Stewart S. Epidemiology, aetiology, and prognosis of heart failure. Heart. 2000 May;83(5):596-602. doi: 10.1136/heart.83.5.596. No abstract available. PMID 10768918
- [Result] Rubler S, Dlugash J, Yuceoglu YZ, Kumral T, Branwood AW, Grishman A. New type of cardiomyopathy associated with diabetic glomerulosclerosis. Am J Cardiol. 1972 Nov 8;30(6):595-602. doi: 10.1016/0002-9149(72)90595-4. No abstract available. PMID 4263660
- [Result] Poornima IG, Parikh P, Shannon RP. Diabetic cardiomyopathy: the search for a unifying hypothesis. Circ Res. 2006 Mar 17;98(5):596-605. doi: 10.1161/01.RES.0000207406.94146.c2. PMID 16543510
- [Result] Fein FS, Strobeck JE, Malhotra A, Scheuer J, Sonnenblick EH. Reversibility of diabetic cardiomyopathy with insulin in rats. Circ Res. 1981 Dec;49(6):1251-61. doi: 10.1161/01.res.49.6.1251. PMID 7030513
- [Result] Hiramatsu K, Ohara N, Shigematsu S, Aizawa T, Ishihara F, Niwa A, Yamada T, Naka M, Momose A, Yoshizawa K. Left ventricular filling abnormalities in non-insulin-dependent diabetes mellitus and improvement by a short-term glycemic control. Am J Cardiol. 1992 Nov 1;70(13):1185-9. doi: 10.1016/0002-9149(92)90053-2. PMID 1414944
- [Result] Iliadis F, Kadoglou N, Didangelos T. Insulin and the heart. Diabetes Res Clin Pract. 2011 Aug;93 Suppl 1:S86-91. doi: 10.1016/S0168-8227(11)70019-5. PMID 21864757
- [Result] Cohen P, Harel C, Bergman R, Daoud D, Pam Z, Barzilai N, Armoni M, Karnieli E. Insulin resistance and acanthosis nigricans: evidence for a postbinding defect in vivo. Metabolism. 1990 Oct;39(10):1006-11. doi: 10.1016/0026-0495(90)90158-9. PMID 2215248
- [Result] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Result] Whitlow PL, Rogers WJ, Smith LR, McDaniel HG, Papapietro SE, Mantle JA, Logic JR, Russell RO Jr, Rackley CE. Enhancement of left ventricular function by glucose-insulin-potassium infusion in acute myocardial infarction. Am J Cardiol. 1982 Mar;49(4):811-20. doi: 10.1016/0002-9149(82)91963-4. No abstract available. PMID 7039286
- [Result] Rizza RA, Mandarino LJ, Gerich JE. Dose-response characteristics for effects of insulin on production and utilization of glucose in man. Am J Physiol. 1981 Jun;240(6):E630-9. doi: 10.1152/ajpendo.1981.240.6.E630. PMID 7018254
- [Result] Cohen P, Barzilai N, Barzilai D, Karnieli E. Correlation between insulin clearance and insulin responsiveness: studies in normal, obese, hyperthyroid, and Cushing's syndrome patients. Metabolism. 1986 Aug;35(8):744-9. doi: 10.1016/0026-0495(86)90242-8. PMID 3526086
- [Result] Khouri SJ, Maly GT, Suh DD, Walsh TE. A practical approach to the echocardiographic evaluation of diastolic function. J Am Soc Echocardiogr. 2004 Mar;17(3):290-7. doi: 10.1016/j.echo.2003.08.012. PMID 14981433
- [Result] Jonassen AK, Sack MN, Mjos OD, Yellon DM. Myocardial protection by insulin at reperfusion requires early administration and is mediated via Akt and p70s6 kinase cell-survival signaling. Circ Res. 2001 Dec 7;89(12):1191-8. doi: 10.1161/hh2401.101385. PMID 11739285
- [Result] Kahn JK, Zola B, Juni JE, Vinik AI. Radionuclide assessment of left ventricular diastolic filling in diabetes mellitus with and without cardiac autonomic neuropathy. J Am Coll Cardiol. 1986 Jun;7(6):1303-9. doi: 10.1016/s0735-1097(86)80150-4. PMID 3011872
- [Result] Sasso FC, Carbonara O, Cozzolino D, Rambaldi P, Mansi L, Torella D, Gentile S, Turco S, Torella R, Salvatore T. Effects of insulin-glucose infusion on left ventricular function at rest and during dynamic exercise in healthy subjects and noninsulin dependent diabetic patients: a radionuclide ventriculographic study. J Am Coll Cardiol. 2000 Jul;36(1):219-26. doi: 10.1016/s0735-1097(00)00717-8. PMID 10898438
- [Result] Khankirawatana B, Khankirawatana S, Peterson B, Mahrous H, Porter TR. Peak atrial systolic mitral annular velocity by Doppler tissue reliably predicts left atrial systolic function. J Am Soc Echocardiogr. 2004 Apr;17(4):353-60. doi: 10.1016/j.echo.2003.12.023. PMID 15044870
- [Result] Mak GS, Sawaya H, Khan AM, Arora P, Martinez A, Ryan A, Ernande L, Newton-Cheh C, Wang TJ, Scherrer-Crosbie M. Effects of subacute dietary salt intake and acute volume expansion on diastolic function in young normotensive individuals. Eur Heart J Cardiovasc Imaging. 2013 Nov;14(11):1092-8. doi: 10.1093/ehjci/jet036. Epub 2013 Mar 20. PMID 23515219
- [Result] Diaz R, Goyal A, Mehta SR, Afzal R, Xavier D, Pais P, Chrolavicius S, Zhu J, Kazmi K, Liu L, Budaj A, Zubaid M, Avezum A, Ruda M, Yusuf S. Glucose-insulin-potassium therapy in patients with ST-segment elevation myocardial infarction. JAMA. 2007 Nov 28;298(20):2399-405. doi: 10.1001/jama.298.20.2399. PMID 18042917
- [Result] Mamas MA, Neyses L, Fath-Ordoubadi F. A meta-analysis of glucose-insulin-potassium therapy for treatment of acute myocardial infarction. Exp Clin Cardiol. 2010 Summer;15(2):e20-4. PMID 20631859
- [Derived] Daoud Naccache D, Yalonetsky S, Bar-Yoseph R. Acute Effects of Insulin on Cardiac Function in Patients with Diabetes Mellitus: Clinical Applicability and Feasibility. Int J Endocrinol. 2020 Mar 17;2020:8134548. doi: 10.1155/2020/8134548. eCollection 2020. PMID 32308680